CLINICAL TRIAL: NCT00567021
Title: German PMS Trial (AWB) to Evaluate Therapy in Reflux Disease and NSAR-Symptoms
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr. Kai Ritcher, AstraZeneca Germany
Other Study IDs: 1312004007; German PMS trial no.7
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Gastroesophageal Reflux
Keywords: reflux; NSAR treatment; Patients with reflux symptoms or gastrointestinal symptoms after NSAR Treatment
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with GERD or NSAID-related ulcers

SUMMARY:
This PMS study had the objective to evaluate under ordinary medical care conditions the efficacy and tolerability of esomeprazole in patients who where treated by general practitioners and internists.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GERD, or NSAID related ulcers, who need treatment with esomeprazole.

Exclusion Criteria:

* Limitations; possible risks; warnings; contraindications mentioned in the SPC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PC and internist
Enrollment: 67130 (Actual)
Dates: Start 2005-09; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To gain further insight into the efficacy of esomeprazole under ordinary medical care conditions in consideration of diagnosis and type of NSAID therapy (if administered). | By estimating the proportion of treated subjects without any gastrointestinal symptoms at the end of the observational period 2. by assessing the change in intensity of gastrointestinal symptoms.

SECONDARY OUTCOMES:
To get further insight into the details of the use, dosage scheme and duration of treatment with esomeprazole in this population

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MD, Study Director — AstraZeneca Medical Department